CLINICAL TRIAL: NCT05538000
Title: Evaluation of the Feasibility of Personalized and Preventive Support for COGnitive Complaints, by a Paramedical Caregiver in Women Suffering From Non-Metastatic Breast Cancer, Requiring Chemotherapy (EFACog).
Brief Title: Personalized Preventive Support for Cognitive Impairment in Non-Metastatic Breast Cancer (EFACog)
Acronym: EFACog
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICL-2022-1
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: No Metastatic Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized support program (Experimental)
  Interventions: Other: Face to face and telephonic interviews

INTERVENTIONS:
Other: Face to face and telephonic interviews — face to face interview : before the first chemotherapy treatment (M0), then at 3 months (M3), 6 months (M6) and 9 months (M9) after the first chemotherapy treatment.
  Telephonic interview : every month between two face-to-face interviews, i.e. at 1 month after the first treatment (M1), at 2 months (M2), at 4 months (M4), at 5 months (M5), at 7 months (M7) and at 8 months (M8) after the first chemotherapy treatment.

SUMMARY:
EFACog is a single-center prospective cohort feasibility study conducted on a single group of patients to study the feasibility of a personalized support program by a nurse conducted over 9 months, using face-to-face and telephone interviews. The objective of this support program is to prevent the occurrence of post-chemotherapy cognitive impairment. After a pre-inclusion visit, patients with no pre-existing cognitive impairment will be included in the study and will receive a 9-month follow-up after the first course of chemotherapy. All follow-up visits (telephone or face-to-face) will be scheduled in conjunction with those taking place in the care setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65;
* WHO 0 to 1;
* Patient newly diagnosed with breast cancer (unilateral or bilateral);
* Patient with a MoCA score not revealing proven cognitive disorders (MoCA ≥ 26/30 and a QPC score <3, without a "YES" answer to question 5 and without 2 "YES" answers to questions A, 4, 5, 7, 8 of the questionnaire);
* Patient to receive adjuvant or neo-adjuvant chemotherapy;
* Patient having understood, signed and dated the consent form
* Affiliated to a social security system

Exclusion Criteria:

* Patient with a cancer concomitant with breast cancer and/or metastatic breast cancer;
* Patients with previous or ongoing carcinological treatment;
* Patient with a major cognitive disorder or a significant cognitive complaint (according to MoCA < 26/30 and QPC >3 with "YES" answer to question 5 and with 2 "YES" answers to questions A, 4, 5, 7, 8 of the questionnaire) or neurological sequelae (epilepsy or neurodegenerative disease);
* Patients who are hearing impaired, visually impaired, or unable to read or speak French
* Patient deprived of liberty (including curatorship and guardianship);
* Pregnant woman;
* Man.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2027-06-17 (Estimated)

PRIMARY OUTCOMES:
To assess program feasibility | 9 months
  Rate of patients who participated in all provider interviews (face-to-face and telephone contacts).

SECONDARY OUTCOMES:
The cognitive complaint | 9 months
  The cognitive complaint will be assessed by the FACT-Cog questionnaire comprising 37 items.
The Quality of life of patients | 9 months
  Quality of life will be assessed by the generic QLQ-C30 questionnaire of 30 items.
Fatigue | 9 months
  Fatigue will be assessed by the QLQ-FA12 questionnaire of 12 items.
Anxiety and depression | 9 months
  Anxiety/depression will be assessed by the 14-item HADS questionnaire (7 items: anxiety / 7 items: depression).
Appearance of neurocognitive disorders and/or significant cognitive complaints | 9 months
  The appearance of neurocognitive disorders and/or significant cognitive complaints will be assessed by taking the MoCA (Montreal Cognitive Assessment) and QPC (Semi-structured Cognitive Complaint Questionnaire) tests.
Satisfaction of patients | 9 months
  Satisfaction will be assessed by a numerical scale (0: not satisfied to 10: very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: LIONEL UWER, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Vandoeuvres Les Nancy, France